CLINICAL TRIAL: NCT04499638
Title: Incidence of Complications of Peripheral Venous Access in the Type 2 Diabetic Population. Analysis of Risk Factors and Comparative Study of Two Peripheral Devices
Brief Title: Incidence of Complications of Peripheral Venous Access in the Type 2 Diabetic Population
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)74/2020
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2; Catheterization, Peripheral; Upper Extremity Deep Vein Thrombosis; Catheter-Related Infections; Diabetes Complications
Keywords: Diabetes Mellitus Type 2; Catheter-Related complications; Short peripheral venous catheter; Medium line peripheral catheter (Midline); Peripheral Insertion Central Catheter (PICC)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Upper Extremity Deep Vein Thrombosis; Catheter-Related Infections; Diabetes Complications | interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non type 2 diabetic patient: Tracking the catheter from insertion to removal. Collection of any patients complication associated with these devices and what different treatments has been administered
  Interventions: Device: Peripheral vascular catheters
- Diabetic type 2 patient: Tracking the catheter from insertion to removal.Collection of any patients complication associated with these devices and what different treatments has been administered
  Interventions: Device: Peripheral vascular catheters

INTERVENTIONS:
Device: Peripheral vascular catheters — Carry time of common peripheral vascular devices in clinical practice and the reason for his withdrawal
  Other Names: Short canula, Midline, PICC

SUMMARY:
Diabetes Mellitus type 2 (T2DM) is one of the most frequent metabolic diseases worldwide. It is expected that in 2035 around 600 million people will suffer from the disease. A recent systematic review has estimated that the direct annual cost of Diabetes worldwide treatments and care is over $ 827 billion and has been independently associated with nosocomial complications, thrombosis-like infections and prolonged admissions. In addition, it is estimated that up to 90% of patients in acute hospitals require a peripheral venous catheter which are associated at the same time with mechanical, infectious and thrombotic acute complications. Recently the emergence of new medium-sized peripheral devices (Midline®) and new peripheral central venous access catheters (PICC), which are more biocompatible, are opening new clinical possibilities with the aim of improving safety and comfort during treatment time and the reduction of associated complications.

With all this, an observational case-control study has been proposed in order to analyse the impact of T2DM disease and its associated complications on the patient requiring peripheral venous access. Furthermore investigators will consider if these new peripheral devices can be a remarkable benefit for these patients. This study will be carried out at the Vall d'Hebron University Hospital in Barcelona, Spain

DETAILED DESCRIPTION:
This Prospective case-control study will be carried out with patients that will be admitted in the hospitalization areas of the Vall d'Hebron Hospital. All research data will be collected by the hospital's vascular access nursing team. Complications related to peripheral venous access (phlebitis, thrombosis, pain, erythema, extravasation) and the time of catheter replacement are the focus outcomes of the present study and possible differences between the control group and the sample population of the T2DM will be analysed. General clinical and anthropometric data (age, sex, BMI, toxic habits,...), cause of admission, co-morbidities, and all variables related to diabetes (time of evolution, degree of glycemic control, treatment, and presence of chronic complications) will also be collected. If there are any significant differences, they will be related to the different risk factors associated with T2DM through association of different epidemiological variables. Furthermore in this hypothetical case, the research team would intend to develop and carry out molecular studies through analysis of blood and urine components, proteinomics and genetic studies.

Hypothesis:

* T2DM is an independent risk factor for catheter-related complications.
* The use of new vascular access devices (Midline, PICC) in patients with T2DM would be associated with a lower risk of catheter-related complications.

Main objective:

- To assess the influence of T2DM on complications related to peripheral vascular catheters in hospitalized patients.

It is expected to colect information of N=500 samples, 250 control group (noT2DM subjects) and 250 study group (T2DM subjects). Due to previous experience, the sample proposed is totally acceptable

ELIGIBILITY:
Inclusion Criteria:

* Peripheral venous access requirement >7 days
* Administration of intravenous treatment

Exclusion Criteria:

* Peripheral venous access for urgent or life-threatening pathology
* Acute psychiatric pathology
* Impossibility of peripheral venous access through the upper limb (amputations, extensive burns, etc.)
* History of venous thrombosis due to catheter less than 1 year

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our hospital who require intravenous treatment and a peripheral venous device has been placed
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
How is the influence of T2DM on complications related to peripheral vascular catheters in hospitalized patients | 12 month
  Rate of complications associated with catheters: thrombosis, infection, pain and skin reaction

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Simó, Prof., Study Director — Vall Hebron Research Institute-VHIR
Locations (1):
- Vall d'Hebron Research Institute-VHIR, Barcelona, Spain

REFERENCES:
- [Background] Nowotny K, Jung T, Hohn A, Weber D, Grune T. Advanced glycation end products and oxidative stress in type 2 diabetes mellitus. Biomolecules. 2015 Mar 16;5(1):194-222. doi: 10.3390/biom5010194. PMID 25786107
- [Background] Asmat U, Abad K, Ismail K. Diabetes mellitus and oxidative stress-A concise review. Saudi Pharm J. 2016 Sep;24(5):547-553. doi: 10.1016/j.jsps.2015.03.013. Epub 2015 Mar 21. PMID 27752226
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2017 Abridged for Primary Care Providers. Clin Diabetes. 2017 Jan;35(1):5-26. doi: 10.2337/cd16-0067. No abstract available. PMID 28144042
- [Background] Tangvarasittichai S. Oxidative stress, insulin resistance, dyslipidemia and type 2 diabetes mellitus. World J Diabetes. 2015 Apr 15;6(3):456-80. doi: 10.4239/wjd.v6.i3.456. PMID 25897356
- [Background] Hurrle S, Hsu WH. The etiology of oxidative stress in insulin resistance. Biomed J. 2017 Oct;40(5):257-262. doi: 10.1016/j.bj.2017.06.007. Epub 2017 Nov 8. PMID 29179880
- [Background] Banerjee M, Vats P. Reactive metabolites and antioxidant gene polymorphisms in Type 2 diabetes mellitus. Redox Biol. 2014;2:170-7. doi: 10.1016/j.redox.2013.12.001. Epub 2013 Dec 11. PMID 25460725
- [Background] Ley SH, Ardisson Korat AV, Sun Q, Tobias DK, Zhang C, Qi L, Willett WC, Manson JE, Hu FB. Contribution of the Nurses' Health Studies to Uncovering Risk Factors for Type 2 Diabetes: Diet, Lifestyle, Biomarkers, and Genetics. Am J Public Health. 2016 Sep;106(9):1624-30. doi: 10.2105/AJPH.2016.303314. Epub 2016 Jul 26. PMID 27459454
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Lowe G, Woodward M, Hillis G, Rumley A, Li Q, Harrap S, Marre M, Hamet P, Patel A, Poulter N, Chalmers J. Circulating inflammatory markers and the risk of vascular complications and mortality in people with type 2 diabetes and cardiovascular disease or risk factors: the ADVANCE study. Diabetes. 2014 Mar;63(3):1115-23. doi: 10.2337/db12-1625. Epub 2013 Nov 12. PMID 24222348
- [Background] Seuring T, Archangelidi O, Suhrcke M. The Economic Costs of Type 2 Diabetes: A Global Systematic Review. Pharmacoeconomics. 2015 Aug;33(8):811-31. doi: 10.1007/s40273-015-0268-9. PMID 25787932
- [Background] Sayampanathan AA. Systematic review of complications and outcomes of diabetic patients with burn trauma. Burns. 2016 Dec;42(8):1644-1651. doi: 10.1016/j.burns.2016.06.023. Epub 2016 Aug 29. PMID 27595452
- [Background] Low ZK, Ng WY, Fook-Chong S, Tan BK, Chong SJ, Hwee J, Tay SM. Comparison of clinical outcomes in diabetic and non-diabetic burns patients in a national burns referral center in Southeast Asia: A 3-year retrospective review; Methodological issues. Burns. 2017 Sep;43(6):1368. doi: 10.1016/j.burns.2017.03.019. Epub 2017 Jun 9. No abstract available. PMID 28602590
- [Background] Vondran M, Schack S, Garbade J, Binner C, Mende M, Rastan AJ, Borger MA, Schroeter T. Evaluation of risk factors for a fulminant Clostridium difficile infection after cardiac surgery: a single-center, retrospective cohort study. BMC Anesthesiol. 2018 Sep 27;18(1):133. doi: 10.1186/s12871-018-0597-2. PMID 30257648
- [Background] Keogh S, Marsh N, Higgins N, Davies K, Rickard C. A time and motion study of peripheral venous catheter flushing practice using manually prepared and prefilled flush syringes. J Infus Nurs. 2014 Mar-Apr;37(2):96-101. doi: 10.1097/NAN.0000000000000024. PMID 24583939
- [Background] Bomberg H, Kubulus C, List F, Albert N, Schmitt K, Graber S, Kessler P, Steinfeldt T, Standl T, Gottschalk A, Wirtz SP, Burgard G, Geiger P, Spies CD, Volk T; German Network for Regional Anaesthesia Investigators. Diabetes: a risk factor for catheter-associated infections. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):16-21. doi: 10.1097/AAP.0000000000000196. PMID 25474624
- [Background] Liem TK, Yanit KE, Moseley SE, Landry GJ, Deloughery TG, Rumwell CA, Mitchell EL, Moneta GL. Peripherally inserted central catheter usage patterns and associated symptomatic upper extremity venous thrombosis. J Vasc Surg. 2012 Mar;55(3):761-7. doi: 10.1016/j.jvs.2011.10.005. PMID 22370026
- [Background] Bahl A, Hang B, Brackney A, Joseph S, Karabon P, Mohammad A, Nnanabu I, Shotkin P. Standard long IV catheters versus extended dwell catheters: A randomized comparison of ultrasound-guided catheter survival. Am J Emerg Med. 2019 Apr;37(4):715-721. doi: 10.1016/j.ajem.2018.07.031. Epub 2018 Jul 19. PMID 30037560
- [Background] Pittiruti M, Brutti A, Celentano D, Pomponi M, Biasucci DG, Annetta MG, Scoppettuolo G. Clinical experience with power-injectable PICCs in intensive care patients. Crit Care. 2012 Feb 4;16(1):R21. doi: 10.1186/cc11181. PMID 22305301
- [Background] Potet J, Arnaud FX, Thome A, Weber-Donat G, Konopacki J, Bouzad C, Kervella Y, Erauso T, Garcia G, Evelyne P, Valbousquet L, Baccialone J, Teriitehau CA. Peripherally inserted central catheter placement in patients with coagulation disorders: A retrospective analysis. Diagn Interv Imaging. 2015 Nov;96(11):1147-51. doi: 10.1016/j.diii.2014.12.012. Epub 2015 May 27. PMID 26025158
- [Background] Gao Y, Fan X, Han J. Prognostic factors for venous thrombosis in patients with peripherally inserted central catheters: Protocol for a systematic review and meta-analysis. Medicine (Baltimore). 2020 Jul 10;99(28):e21037. doi: 10.1097/MD.0000000000021037. PMID 32664112
- [Background] Miliani K, Taravella R, Thillard D, Chauvin V, Martin E, Edouard S, Astagneau P; CATHEVAL Study Group. Peripheral Venous Catheter-Related Adverse Events: Evaluation from a Multicentre Epidemiological Study in France (the CATHEVAL Project). PLoS One. 2017 Jan 3;12(1):e0168637. doi: 10.1371/journal.pone.0168637. eCollection 2017. PMID 28045921